CLINICAL TRIAL: NCT00578422
Title: Clinical Implications of Peripheral Plaque Morphology
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 6723; 5R01HL075721-05 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Peripheral Artery Disease
Keywords: PAD; Peripheral Artery Disease; IVUS; Plaque
MeSH Terms: conditions — Peripheral Arterial Disease; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm I: In Vitro IVUS Plaque studies: IVUS of Amputation Specimens
  Interventions: Other: Ivus (Intravascular Ultrasound) of Amputation Specimens
- Arm 2: Obserational Study: IVUS for patients undergoing standard lower extremity angiography for PAD.
  Interventions: Procedure: IVUS (Intravascular Ultrasound)

INTERVENTIONS:
Other: Ivus (Intravascular Ultrasound) of Amputation Specimens — Human lower extremity arterial segments will be obtained at autopsy and from amputation specimens. All imaging studies and vessel fixation will be undertaken immediately upon vessel procurement; in most cases this will occur within 2 hours of dissection and within 24 hours of death. The ex vivo portion of the study will make use of 150 excised vessels obtained over a 48-month period from randomly selected autopsy cases. From these vessels we expect to collect data from a minimum of 560 plaques
  Groups: Arm I: In Vitro IVUS Plaque studies
Procedure: IVUS (Intravascular Ultrasound) — Standard diagnostic arteriographic images will be obtained. Appropriate oblique views will be acquired at the common femoral bifurcation. Next, IVUS will be performed obtaining ultrasound data from a 10 cm lower extremity artery.
  Groups: Arm 2: Obserational Study

SUMMARY:
Peripheral Artery Disease involves a buildup of fatty deposits (plaque) within blood vessels that can restrict blood flow. Patients who have PAD and claudication (pain in legs during exercise due to poor blood circulation) may be eligible for this clinical trial. Three primary hypotheses will be tested in this study: (1) IVUS (Intravascular Ultrasound)combined with advanced digital image and signal processing provides a sensitive method to determine plaque geometry and composition in the human peripheral artery wall; (2) IVUS can discern specific arterial wall morphology, providing data that can be used to identify plaques that predispose the patient to late complications; and (3) IVUS-derived plaque structure can be used to predict responders and non-responders to pharmacologic therapy and percutaneous endovascular interventions. These hypotheses will be tested as follows: (1) custom engineered IVUS analysis software will be used to describe the geometry, composition, and spatial component relationships of the vessel, (2) the morphology of lower extremity arterial plaque, as determined by IVUS, will be correlated with baseline clinical characteristics of subjects, and (3) the effects on plaque morphology after long term treatment with antihyperlipidemics will be determined.

DETAILED DESCRIPTION:
Advances in the pathophysiology of Peripheral Arterial Disease (PAD) have been limited by the inaccessibility of the blood vessels to precise diagnostic interrogation. Traditional methods for studying disease in the peripheral arterial blood vessels have significant limitations. The development and refinement of IVUS (Intravascular Ultrasound) has provided a powerful in vivo method to assess plaque morphology. The potential of IVUS to quantify the structure and geometry of normal and atherosclerotic peripheral arteries will allow one to characterize specific lesions and to distinguish which plaques will or will not lead to complications.

Three primary hypotheses will be tested in this study: (1) IVUS combined with advanced digital image and signal processing provides a sensitive method to determine plaque geometry and composition in the human peripheral artery wall; (2) IVUS can discern specific arterial wall morphology, providing data that can be used to identify plaques that predispose the patient to late complications; and (3) IVUS-derived plaque structure can be used to predict responders and non-responders to pharmacologic therapy and percutaneous endovascular interventions.

These hypotheses will be tested as follows: (1) custom engineered IVUS analysis software will be used to describe the geometry, composition, and spatial component relationships of the vessel, (2) the morphology of lower extremity arterial plaque, as determined by IVUS, will be correlated with baseline clinical characteristics of subjects, and (3) the effects on plaque morphology after long term treatment with antihyperlipidemics will be determined.

There are three arms of the trial. (1) IVUS of Amputation Specimens: Histological sections of fresh arterial segments from amputation specimens will be correlated with IVUS derived radiofrequency data to quantify arterial plaque burden and composition (dense calcium, fibrous, fibro-fatty, and necrotic core components). (2)Observational Study: Patients undergoing standard lower extremity angiography for PAD will be studied with IVUS at the same sitting. IVUS finding will be correlated with demographic factors (age, gender, and race) and symptom severity (claudication, rest pain, tissue loss). Patients will be followed up for up to five years, and the occurrence of ischemic events (worsening of leg ischemia, need for intervention and re-intervention, and distant complications such as MI and stroke) will be reconciled with the arterial wall at the baseline examination. (3) Randomized Clinical Trial: A randomized, double-blinded clinical trial of high-dose atorvastatin vs. low dose atorvastatin will be performed in patients with intermittent claudication, based on our hypothesis with statin therapy will result in stabilization or regression of lower extremity arterial plaque, differences best assessed with high resolution imaging studies. Enrollment goals were not met due to treatment paradigm that has shifted to aggressive LDL control, therefore the overwhelming majority of patients were excluded due their existing statin therapy. On 6/25/08 the protocol and informed consent were amended to reflect elimination of the Randomized arm of this study and the restructuring of this arm to a Cohort Observational arm, correlating patients' current statin dosages with LDL levels and plaque morphology. This is the current design for this arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Symptoms of intermittent claudication, rest pain, or minor tissue loss (Rutherford Category I - V).99
3. Non invasive laboratory evidence of peripheral vascular disease.
4. Angiographic demonstration of a 100 mm patent segment of a lower extremity artery containing at least one visually estimated stenosis of 20 - 80% diameter reduction.

Exclusion Criteria:

1. Acute limb ischemia, defined by a significant change in symptoms (one category on the Rutherford scale99 within the previous 14 days).
2. Concurrent oral anticoagulant therapy that cannot be safely withheld.
3. Extensive tissue loss and/or gangrene which would result in an above knee or below knee amputation(s).

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PAD undergoing standard lower extremity angiography.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2003-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Develop automated algorithms to determine plaque geometry and composition from IVUS "backscattered" data | within 24 hours of amputation
  Spectral analysis of plaque

SECONDARY OUTCOMES:
Clinical Correlation: Plaque Structure and Composition | During angiography for PAD
  IVUS concurrent with angiography

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Eagleton, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No